CLINICAL TRIAL: NCT01485848
Title: EP-100, a Novel LHRH Receptor-Targeted, Membrane-Disrupting Peptide, Plus Paclitaxel Versus Paclitaxel Alone for Refractory or Recurrent Ovarian Cancer: A Phase II, Randomized, Multicenter Trial
Brief Title: EP-100 Plus Paclitaxel Versus Paclitaxel Alone in Patients With Ovarian Cancer
Acronym: ESP2011-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperance Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT12601; U1111-1124-2062 (Other: UTN)
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — EP-100 membrane-disrupting peptide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel (Active Comparator): A single 1 hour intravenous infusion every week for 6 cycles (each cycle is 4 weeks)
  Interventions: Drug: EP-100
- Paclitaxel + EP-100 (Experimental): Paclitaxel every week plus EP-100 twice weekly by 1 hour intravenous infusion for the first 3 weeks of each 4 week cycle for 6 cycles (each cycle is 4 weeks)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: EP-100 — Pharmaceutical form:Solution Route of administration: Intravenous
  Arms: Paclitaxel
Drug: Paclitaxel — Pharmaceutical form:Solution Route of administration: Intravenous
  Arms: Paclitaxel + EP-100

SUMMARY:
Primary Objectives: o Run-in Phase: Determine a dose of EP-100 at which the initial benefit/risk of paclitaxel combined with EP-100 can be studied. o Randomized Phase: Compare the anti-tumor effects of EP-100 combined with weekly paclitaxel versus paclitaxel alone in patients with ovarian cancer. Secondary Objectives: o Randomized Phase: Quantify any significant changes in the safety profile of weekly paclitaxel alone compared to the doublet combination of paclitaxel with EP-100. o Determine an initial benefit/risk profile for this new drug combination.

DETAILED DESCRIPTION:
Total duration of the study for each participant is 9 to 10 months, consisting of a 1 month screening period, a 6 to 7 months treatment period, and a 30 day follow-up. All patients with stable disease or who have achieved partial or complete response and for whom dosing has been safe and reasonably well-tolerated may continue additional treatment cycles on the same regimen. Any patient whose imaging assessment shows disease progression after receiving at least two cycles of single agent weekly paclitaxel on ARM 1 may then be offered treatment with the combination of EP-100 plus paclitaxel in the same dose regimen as ARM 2.

ELIGIBILITY:
Inclusion criteria:

* Adult patients with histologically confirmed epithelial ovarian carcinomas; these will include primary peritoneal and fallopian tube carcinomas. Patient's tumor shown to be positive for the LHRH-receptors by standardized immunocytochemistry performed at the study's central laboratory.
* Reliable cancer treatment history documenting advanced disease in patients who have progressed during or recurred after treatment with a paclitaxel and/or platinum regimen for advanced disease.
* Evaluable disease based on criteria of the Gynecologic Intergroup Response Evaluation Criteria in in Solid Tumors.
* Karnofsky performance status >/= 70%.

Exclusion criteria:

* Significant cardiac disease.
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
* Pregnant or nursing women.
* Treatment with radiation therapy or investigational therapy within 4 weeks prior to Day 1. Had received chemotherapy prior to study entry equivalent to 3 to 5 half-lives of that chemotherapy agent or 4 weeks prior to study entry (whichever is shorter) with resolution of any side effects from that previous therapy (6 weeks for nitrosoureas or Mitomycin C.)
* Subjects with known central nervous system (CNS) metastases, either previously treated or current.
* Disease-free and off therapy for any other cancer within 5 years, except for adequately treated basal cell or squamous cell skin cancer or cervical intraepithelial neoplasia (CIN).
* Had major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1. o Had minor surgery (superficial incisions unlikely to obscure bleeding or infections) within 2 weeks prior to Day 1.
* Potentially life-threatening disease (hypercalcemia, spinal cord compression) whose disease may progress acutely during therapy.
* Unwilling or unable to comply with procedures required in this protocol.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Susceptibility to histamine release.
* Chronic treatment with corticosteroids.
* Baseline QTc exceeding 450 msec (by Bazett's formula) and/or patients receiving class 1A or class III antiarrythmic agents.
* Serious nonmalignant disease.
* Subjects who are currently receiving any other investigational agent.
* Inadequate renal and liver functions and bone marrow reserve.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities (DLTs) at different doses | Up to 30 weeks
Overall Response Rate (ORR) | Up to 30 weeks

SECONDARY OUTCOMES:
Time to Progression (TTP) - Time | Up to 18 months
Progression-free Survival - Time | Up to 18 months
Overall Survival (OS) - Time | Up to 18 months
Duration of Response - Time | Up to 18 months
Number of Participants with Adverse Events | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Investigational Site Number 840001, Greenbrae, California
  - Investigational Site Number 840005, San Francisco, California
  - Investigational Site Number 840007, Louisville, Kentucky
  - Investigational Site Number 840010, Covington, Louisiana
  - Investigational Site Number 840011, Shreveport, Louisiana
  - Investigational Site Number 840503, Bozeman, Montana
  - Investigational Site Number 840004, Middletown, Ohio
  - Investigational Site Number 840008, Portland, Oregon
  - Investigational Site Number 840006, Houston, Texas
  - Investigational Site Number 840603, Kennewick, Washington
  - Investigational Site Number 840103, Mount Vernon, Washington
  - Investigational Site Number 840403, Seattle, Washington
  - Investigational Site Number 840003, Seattle, Washington
  - Investigational Site Number 840303, Tacoma, Washington
  - Investigational Site Number 840203, Wenatchee, Washington